CLINICAL TRIAL: NCT02061852
Title: Prospective Trial for the Evaluation of Safety, Tolerability and Efficacy of the Medical Device Simeox ® Compared to Traditional Respiratory Physiotherapy Techniques for Airway Secretion Clearance
Brief Title: Evaluation of the Safety of the Medical Device Simeox®
Acronym: SIMETOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Physio-Assist (Industry)
Collaborators: CEISO (Industry); University Hospital, Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00079-38
Record Dates: First submitted 2014-01-31; First posted 2014-02-13 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Broncho-degenerative Disease; Chronic Obstructive Airway Disease; Cystic Fibrosis; Idiopathic Bronchiectasis; Ciliary Dyskinesia; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis; Ciliary Motility Disorders; Bronchitis, Chronic | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy (Active Comparator): Traditional techniques
  Interventions: Device: Simeox; Procedure: Physiotherapy
- simeox (Experimental): Medical device
  Interventions: Device: Simeox; Procedure: Physiotherapy

INTERVENTIONS:
Device: Simeox
Procedure: Physiotherapy

SUMMARY:
The purpose of this study is to determine whether the medical device "simeox" is safe in the treatment of respiratory diseases, in comparison with traditional physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18, male or female.
* Patient affected by broncho-degenerative disease, chronic obstructive airway disease, cystic fibrosis, idiopathic bronchiectasis, ciliary dyskinesia and/or chronic bronchitis.
* Hospitalization for a minimum of five days or a maximum of 8 days.
* Bronchial clearance is usually productive.
* FVC and / or FEV <85% predicted, with stable lung function.
* Agreement to participate to the study and signature of the informed consent form
* Social security coverage.

Exclusion Criteria:

* Patient infected with bacteria resistant to antibiotics.
* Bronchial clearance is not usually productive.
* Patient with contra-indication for physiotherapy bronchial clearance.
* Patient who received a lung transplant.
* Care requires more than 2 sessions of chest physiotherapy daily.
* Duration of mechanical ventilation > 8h/day.
* Patient with an episode of hemoptysis during the month before inclusion.
* Patient with an episode of pneumothorax during the last month.
* Pregnant or lactating women.
* Patient with a disability and/or unwillingness to follow protocol requirements.
* Patient participating in another clinical study or having tested an experimental drug within 30 days prior to his inclusion in the study.
* Patient ( s) with another condition which, according to the investigator , may interfere with the result or conduct of the trial and thus justify their non- inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety of the simeox® | Day 8
  Adverse events related or not to the simeox®

CONTACTS AND LOCATIONS:
Overall Officials: Martine Reynaud-Gaubert, Prof., Principal Investigator — Hospital Marseille
Locations (1):
- CHU Nord, Marseille, France